CLINICAL TRIAL: NCT00802763
Title: Performance Proof of the New NORMA-SENSE Panty Liner - in-Vivo STUD
Brief Title: Performance Proof of the New NORMA-SENSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: common sense, COMMON SENSE
Other Study IDs: F-7-28.1-1 VER-2
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Vaginal Infection
Keywords: VAGINAL INFECTION; COLOR APPEARANCE; ELEVATED Ph
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — VAGINAL SECRETIONS
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vaginitis
  Interventions: Device: NORMA-SENSE

INTERVENTIONS:
Device: NORMA-SENSE — Should be used by the clinician. the test usage will take up to 6 hours. The result reading will take few second.

SUMMARY:
This study was designed to validate the color appearance on the newly developed panty liner (NORMA-SENSE). The NORMA-SENSE liner changes color when worn by the user and comes into contact with vaginal secretion with an elevated pH level, without false positives due to urine remains or incontinence. The study will also asses the physical comfort in using NORMA-SENSE and the result reading clarity which includes the ability to visualize and interpret the NORMA-SENSE strip results.

ELIGIBILITY:
Inclusion Criteria:

1. Women, age 18 years or greater without symptoms of vaginal infection.
2. Subject is ready to sign the informed consent form.

Exclusion Criteria:

1. Subject is unable or unwilling to cooperate with study procedures.
2. Subject is currently participating in another clinical study.
3. Subject suffers from vaginal bleeding or is menstruating.
4. Subject that have had sexual relations within the last 12 hours.
5. Subject that applied local antiseptic or antibiotic or vaginal treatment within the last 3 days.
6. Subject that applied vaginal douching within 12 hours prior to the visit at the clinic.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women, age greater then 18 without symptoms of vaginal infection.
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
We will asses agreement between the color status of the NORMA-SENSE as reported by the subject after using the panty liner, and the pH measurement with Nitrazine paper. | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Medical center, Haifa, Israel